CLINICAL TRIAL: NCT02630693
Title: Randomized Phase II Study Comparing Two Different Schedules of Palbociclib Plus Second Line Endocrine Therapy in Women With Estrogen Receptor Positive, HER2 Negative Advanced/Metastatic Breast Cancer
Brief Title: Two Different Schedules of Palbociclib + Second Line Endocrine Therapy in Estrogen Receptor Positive, HER2 Neg Advanced/Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA38
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant; Tamoxifen; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palbociclib (100mg) (Active Comparator): Palbociclib 100mg PO daily plus Fulvestrant or Tamoxifen or another Aromatase Inhibitor at the standard doses/schedules
  Interventions: Drug: Palbociclib 100mg; Drug: Fulvestrant or Tamoxifen or Aromatase Inhibitor
- Palbociclib (125mg) (Active Comparator): Palbociclib 125mg PO daily 3 out of 4 weeks plus Fulvestrant or Tamoxifen or another Aromatase Inhibitor at the standard doses/schedules
  Interventions: Drug: Palbociclib 125mg; Drug: Fulvestrant or Tamoxifen or Aromatase Inhibitor

INTERVENTIONS:
Drug: Palbociclib 100mg — 100mg PO daily
  Arms: Palbociclib (100mg)
Drug: Palbociclib 125mg — 125mg PO daily 3 weeks out of 4
  Arms: Palbociclib (125mg)
Drug: Fulvestrant or Tamoxifen or Aromatase Inhibitor — given at the standard doses/schedules

SUMMARY:
The purpose of this study is to determine if the combination of endocrine therapy and Palbociclib at a daily dose of 100 mg will result in a better response to therapy with fewer dose interruptions than the proposed dosing regimen of 125 mg daily for 21 days out of a 28 day cycle in combination with endocrine therapy.

DETAILED DESCRIPTION:
The standard or usual treatment of this type of breast cancer is endocrine therapy. Palbociclib is a new type of drug for breast cancer. Laboratory tests as well as studies in animals and people show that it may help slow the growth of breast cancer. The most widely tested regimen of Palbociclib for patients with metastatic/advanced breast cancer is 125 mg every day for 21 days out of a 28 day cycle in combination with standard endocrine (hormone) therapy. This study explores if administering a lower dose of palbociclib - 100 mg given every day of a 28 day cycle in combination with standard endocrine (hormone) therapy - may result in more tumour shrinkage and be better tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal and postmenopausal women 18 years of age or older.
* Histologically confirmed adenocarcinoma of the breast, with ER positive and HER2 negative status based on local testing on most recent pathological tumour specimen.
* Patients must satisfy the following criteria for prior therapy:

  * Progressed during treatment or within 12 months of completion of adjuvant endocrine therapy or
  * Progressed during prior endocrine therapy for advanced/metastatic disease. Note: 'Progressed during endocrine therapy' means that the patient progressed while on or within 1 month after discontinuation of endocrine therapy.
* One line of chemotherapy for advanced/metastatic disease (regardless of prior adjuvant chemotherapy use) is allowed in addition to endocrine therapy.
* Patients must have evidence of disease to be eligible for the study, but measurable disease is not mandatory.
* For those patient with measureable disease who will be included in the response assessment, the following criteria must apply:

  * X-ray ≥ 20 mm
  * Spiral CT scan or physical exam ≥ 10 mm (lymph nodes must be ≥ 15 mm in the short axis)
  * Conventional CT scan, MRI ≥ 20 mm
  * Measurable lesions must be outside a previous radiotherapy field if they are the sole site of disease, unless disease progression has been documented.

Tumor lesions previously irradiated or subjected to other loco regional therapy will only be deemed measurable if progression at the treated site after completion of therapy is clearly documented.

* Eastern Cooperative Oncology Group (ECOG) 0-2.
* Adequate organ and bone marrow function as defined by:

  * ANC ≥ 1,500/mm3 (1.5 x 109/L)
  * Platelets ≥ 100,000/mm3 (100 x 109/L)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥60 ml/min as calculated using the method standard for the institution;
  * Total serum bilirubin ≤ 1.5 x ULN (<3 ULN if Gilbert's disease).
* Patient must agree to provide tumour tissue from the most recent pathological tumour specimen.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits placed on patients being considered for this trial.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* Women of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Patients with advanced, symptomatic, visceral spread that are at risk of life threatening complication in the short term.
* Patients with symptomatic CNS involvement, meningeal or parenchymal, that is uncontrolled or requires steroids.
* Prior treatment with any CDK 4/6 inhibitor.
* Prior treatment with mTOR inhibitors.
* Active second malignancy, regardless of ongoing treatment.
* Any concurrent medical condition that in the opinion of the investigator would interfere with the safe administration of the study drug and participation in the study.
* Participation in a prior anti-cancer investigational study within 30 days prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil A. Joy, Study Chair — Cross Cancer Institute, Edmonton Alberta Canada
Locations (22):
- Canada (22):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - University Health Network, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy.
URL: https://www.ctg.queensu.ca/public/policies

REFERENCES:
- [Result] Joy AA, Cheng N, Gelmon KA, Mates M, Desbiens C, Clemons M, Taylor S, Lemieux J, DeLuca A, Gasparini L, Lungu I, Soave D, Fortuna A, Pugh T, Liu SS, Bartlett JMS, Awadalla P, Spears M, Chen BE, Bayani J, Parulekar WR. Continuous versus Standard Palbociclib Treatment and Molecular Profiling of Solid Tissues and Liquid Biopsies in the CCTG MA.38 Trial in Advanced Breast Cancer. Cancer Res Commun. 2025 Nov 1;5(11):1998-2011. doi: 10.1158/2767-9764.CRC-25-0346. PMID 41123599
- See also: Related Info — https://doi.org/10.1158/2767-9764.CRC-25-0346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
Started | 90 | 90
Completed | 90 | 89
Not Completed | 0 | 1
Not completed — No receive treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline variables were reported using intend to treat principle
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg) | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 60 | 112
  >=65 years | 38 | 30 | 68
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [53 to 69] | 59.5 [53 to 69] | 60.5 [53 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 90 | 180
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 76 | 75 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 90 | 90 | 180
Menopausal Status [Count of Participants; unit: Participants]
  Postmenopausal | 83 | 80 | 163
  Premenopausal | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Using the RECIST 1.1 Criteria
Description: progression free survival (PFS) is defined as time from randomization to progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Population: Intend to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
Number analyzed (Participants) | 90 | 90
months | 9.33 [6.93 to 13.90] | 11.30 [8.08 to 13.83]
Statistical Analysis 1: Comparison: Palbociclib (100mg) vs Palbociclib (125mg); Test type: Other — As stated in the protocol, the primary objective of this trial is to estimate the hazard ratio and the corresponding 90% confidence interval. Therefore, we do not conduct any statistical hypothesis test for progression free survival; Hazard Ratio (HR) = 0.93, 90% CI 2-sided [0.66 to 1.30] — Hazard ratio of Palbociclib100mg arm vs 125 mg arm

2. Secondary Outcome: Number of Participants With Response or No Response
Description: Response rate = Number of (Complete response + partial response) / total treated patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: Only patients received protocol treatment were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
Number analyzed (Participants) | 90 | 89
Participants
  Response | 10 | 11
  No response | 80 | 78

3. Secondary Outcome: Duration of Response
Description: For patients with complete or partial response, duration of response is defined as days from first recorded response to the first date of recurrent or progression or death.
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
Number analyzed (Participants) | 10 | 11
days | 126 [88 to 251] | 169 [82 to 310]

4. Secondary Outcome: Overall Survival
Description: Time from randomization to death of any cause.
Time Frame: 2 years
Population: Intend to treat population
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
Number analyzed (Participants) | 90 | 90
months | 20.73 [19.29 to 23.30] | 21.39 [19.65 to 26.68]
Statistical Analysis 1: Comparison: Palbociclib (100mg) vs Palbociclib (125mg); Test type: Other — As stated in the protocol, the objective of this trial is to estimate the hazard ratio and the corresponding 90% confidence interval. Therefore, we do not conduct any statistical hypothesis test for overall survival; Hazard Ratio (HR) = 1.07, 90% CI 2-sided [0.67 to 1.69] — Hazard ratio for Palbociclib 100mg arm vs 125 mg arm

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Palbociclib (100mg) | Palbociclib (125mg)
All-Cause Mortality (participants affected / at risk) | 29/90 | 32/89
Serious Adverse Events (participants affected / at risk) | 9/90 | 12/89
Other Adverse Events (participants affected / at risk) | 89/90 | 88/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib (100mg) (N=90) | Palbociclib (125mg) (N=89)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Other general disorders, administration site conditions (General disorders) | 0 (0) | 1 (1)
Other hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib (100mg) (N=90) | Palbociclib (125mg) (N=89)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (5)
Hypothyroidism (Endocrine disorders) | 4 (4) | 5 (5)
Blurred vision (Eye disorders) | 10 (10) | 7 (7)
Dry eye (Eye disorders) | 7 (7) | 4 (4)
Other eye disorders (Eye disorders) | 4 (4) | 9 (9)
Watering eyes (Eye disorders) | 10 (10) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 17 (17) | 22 (22)
Bloating (Gastrointestinal disorders) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 42 (42) | 39 (39)
Diarrhea (Gastrointestinal disorders) | 41 (41) | 37 (37)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 7 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 21 (21) | 22 (22)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 6 (6)
Mucositis oral (Gastrointestinal disorders) | 23 (23) | 24 (24)
Nausea (Gastrointestinal disorders) | 47 (47) | 48 (48)
Oral pain (Gastrointestinal disorders) | 4 (4) | 5 (5)
Other gastrointestinal disorders (Gastrointestinal disorders) | 5 (5) | 4 (4)
Toothache (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 26 (26) | 23 (23)
Chills (General disorders) | 6 (6) | 9 (9)
Edema limbs (General disorders) | 13 (13) | 19 (19)
Fatigue (General disorders) | 77 (77) | 73 (73)
Fever (General disorders) | 11 (11) | 9 (9)
Flu like symptoms (General disorders) | 22 (22) | 11 (11)
Non-cardiac chest pain (General disorders) | 1 (1) | 5 (5)
Pain (General disorders) | 23 (23) | 19 (19)
Allergic reaction (Immune system disorders) | 5 (5) | 3 (3)
Lung infection (Infections and infestations) | 8 (8) | 3 (3)
Other infections and infestations (Infections and infestations) | 5 (5) | 6 (6)
Sinusitis (Infections and infestations) | 7 (7) | 4 (4)
Skin infection (Infections and infestations) | 10 (10) | 4 (4)
Upper respiratory infection (Infections and infestations) | 18 (18) | 23 (23)
Urinary tract infection (Infections and infestations) | 13 (13) | 7 (7)
Wound infection (Infections and infestations) | 5 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Fracture (Injury, poisoning and procedural complications) | 9 (9) | 1 (1)
Weight loss (Investigations) | 6 (6) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 38 (38) | 25 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 33 (33)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (27) | 41 (41)
Bone pain (Musculoskeletal and connective tissue disorders) | 37 (37) | 28 (28)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 21 (21)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 21 (21) | 16 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (38) | 29 (29)
Dizziness (Nervous system disorders) | 17 (17) | 13 (13)
Dysgeusia (Nervous system disorders) | 18 (18) | 13 (13)
Headache (Nervous system disorders) | 34 (34) | 32 (32)
Memory impairment (Nervous system disorders) | 7 (7) | 3 (3)
Other nervous system disorders (Nervous system disorders) | 6 (6) | 3 (3)
Paresthesia (Nervous system disorders) | 13 (13) | 12 (12)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 27 (27) | 30 (30)
Anxiety (Psychiatric disorders) | 25 (25) | 32 (32)
Confusion (Psychiatric disorders) | 5 (5) | 3 (3)
Depression (Psychiatric disorders) | 8 (8) | 24 (24)
Insomnia (Psychiatric disorders) | 44 (44) | 35 (35)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 8 (8)
Breast pain (Reproductive system and breast disorders) | 5 (5) | 9 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 28 (28)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 (40) | 34 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 14 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 32 (32) | 24 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (13) | 9 (9)
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 20 (20) | 18 (18)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 10 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (18) | 20 (20)
Hot flashes (Vascular disorders) | 25 (25) | 39 (39)
Hypertension (Vascular disorders) | 23 (23) | 25 (25)
Lymphedema (Vascular disorders) | 5 (5) | 6 (6)
Thromboembolic event (Vascular disorders) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02630693/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02630693/SAP_001.pdf